CLINICAL TRIAL: NCT01845402
Title: The Prevalence of Chronic Kidney Disease at Adolescence in Patients With Congenital Cardiac Disease, Having Undergone Corrective Surgery During Childhood
Brief Title: Chronic Kidney Disease in Teenagers With Congenital Cardiac Disease
Acronym: PRECARDIO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: P091125
Record Dates: First submitted 2012-12-11; First posted 2013-05-03 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Failure; Congenital Heart Defects
Keywords: Kidney Failure, Chronic; Adolescent; Heart Defects, Congenital
MeSH Terms: conditions — Kidney Failure, Chronic; Heart Defects, Congenital | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sample of blood and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- congenital cardiac diseases: blood sample and urine sample.
  Interventions: Biological: blood and urine samples

INTERVENTIONS:
Biological: blood and urine samples — A blood sample and urine sample will be collected for purpose of the study. CKD (Chronic kidney injury) will be diagnosed according to the KDIGO criteria in children.

SUMMARY:
The prevalence of chronic kidney injury (CKD) following cardiac surgery during childhood is not known, but there is evidence of CKD in young adults. In the present study assumption is made that CKD can already by diagnosed in patients at or just before adolescence, and the aim is calculate its prevalence according to the KDIGO criteria by a cross-sectional study, which will enroll patients aged 10 to 15 years. The second hypothesis is that events occurring peri-operatively during initial surgery or during follow-up could by chart review and regression analysis.

DETAILED DESCRIPTION:
Background. Acute kidney injury is a common complication of cardiac surgery in children. The prevalence of chronic kidney injury (CKD) following cardiac surgery during childhood is not known. The only study published to date is that of Dimopoulos et al., who has estimated the prevalence of CKD in young adults with congenital cardiac diseases at 40% and the prevalence of stage 2 CKD at 6% (Dimopoulos, Circulation 2008). The study by Dimopoulos et al. also showed that CKD was a risk factor of death in this population. Objectives. In the present study assumption is made that CKD can already by diagnosed in patients at or just before adolescence, and the aim is calculate its prevalence. The second hypothesis is that events occurring peri-operatively during initial surgery or during follow-up could be predictive of CKD.

Methodology. The study has been approved by the Ethical Committee of our institution, and is founded by the Departement de la Recherche Clinique et du Developpement, AP-HP, Paris This is a prospective observational cross-sectional study which will enroll patients 10 to 15 years with congenital cardiac diseases, who have undergone surgical repair during childhood. Only patients who have undergone surgery and follow-up at our institution will be enrolled, to insure complete data. The patients will receive complete information about the study by mail that will be send home prior to the appointment for the cardiologic follow-up. After parental and patient consent, a sample of blood and urine will be collected for purpose of the study. CKD will be diagnosed according to the KDIGO criteria in children (Hogg, Pediatrics 2003). In case of CKD, patients will be informed and given an appointment for nephrological support and follow-up at our institution. The prevalence and stage of CKD will be calculated after completion of inclusions. The risk factors of CKD will be identified retrospectively by chart review and regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 10 to15 years, having undergone surgery for congenital heart disease during childhood, and cardiologic follow-up at Necker-Enfants Malades Hospital
* Written informed consent by one parent
* Health insurance

Exclusion Criteria:

* Documented chronic kidney disease of non cardiac origin
* Documented kidney or urinary malformation
* Failure to puncture a peripheral vein

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients 10 to 15 years old with congenital cardiac diseases
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-04-02 (Actual); Primary Completion 2015-06-19 (Actual); Study Completion 2015-06-20 (Actual)

PRIMARY OUTCOMES:
Chronic kidney disease | at Day 0
  The primary measure is the prevalence of chronic kidney disease in teenagers and pre-teenagers with congenital heart disease operated during childhood. For screening purposes, a blood and a urine sample will be collected the day of consultation for the cardiologic follow-up.

SECONDARY OUTCOMES:
Peri-operative risk factors | at day 0
  The secondary aim is the identification of peri-operative risk factors of chronic kidney disease in this population, by retrospective chart-review and regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Mirela Bojan, MD, Principal Investigator — Necker - Enfants Malades Hospital
Locations (1):
- Necker - Enfants Malades Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dimopoulos K, Diller GP, Koltsida E, Pijuan-Domenech A, Papadopoulou SA, Babu-Narayan SV, Salukhe TV, Piepoli MF, Poole-Wilson PA, Best N, Francis DP, Gatzoulis MA. Prevalence, predictors, and prognostic value of renal dysfunction in adults with congenital heart disease. Circulation. 2008 May 6;117(18):2320-8. doi: 10.1161/CIRCULATIONAHA.107.734921. Epub 2008 Apr 28. PMID 18443238
- [Background] Hogg RJ, Furth S, Lemley KV, Portman R, Schwartz GJ, Coresh J, Balk E, Lau J, Levin A, Kausz AT, Eknoyan G, Levey AS; National Kidney Foundation's Kidney Disease Outcomes Quality Initiative. National Kidney Foundation's Kidney Disease Outcomes Quality Initiative clinical practice guidelines for chronic kidney disease in children and adolescents: evaluation, classification, and stratification. Pediatrics. 2003 Jun;111(6 Pt 1):1416-21. doi: 10.1542/peds.111.6.1416. PMID 12777562
- [Background] Levey AS, Eckardt KU, Tsukamoto Y, Levin A, Coresh J, Rossert J, De Zeeuw D, Hostetter TH, Lameire N, Eknoyan G. Definition and classification of chronic kidney disease: a position statement from Kidney Disease: Improving Global Outcomes (KDIGO). Kidney Int. 2005 Jun;67(6):2089-100. doi: 10.1111/j.1523-1755.2005.00365.x. PMID 15882252
- [Background] Pedersen KR, Hjortdal VE, Christensen S, Pedersen J, Hjortholm K, Larsen SH, Povlsen JV. Clinical outcome in children with acute renal failure treated with peritoneal dialysis after surgery for congenital heart disease. Kidney Int Suppl. 2008 Apr;(108):S81-6. doi: 10.1038/sj.ki.5002607. PMID 18379554
- [Background] Askenazi DJ, Feig DI, Graham NM, Hui-Stickle S, Goldstein SL. 3-5 year longitudinal follow-up of pediatric patients after acute renal failure. Kidney Int. 2006 Jan;69(1):184-9. doi: 10.1038/sj.ki.5000032. PMID 16374442
- [Result] Lorut C, Lefebvre A, Planquette B, Quinquis L, Clavier H, Santelmo N, Hanna HA, Bellenot F, Regnard JF, Riquet M, Magdeleinat P, Meyer G, Roche N, Huchon G, Coste J, Rabbat A. Early postoperative prophylactic noninvasive ventilation after major lung resection in COPD patients: a randomized controlled trial. Intensive Care Med. 2014 Feb;40(2):220-227. doi: 10.1007/s00134-013-3150-2. Epub 2013 Nov 29. PMID 24292873